CLINICAL TRIAL: NCT00652288
Title: Evaluation of Pharmacokinetic and Pharmacodynamic Properties of Rapid-Acting Insulin Analogs Given as a Bolus by Continuous Subcutaneous Insulin Infusion (CSII) and in MDI Basal-Bolus Therapy in Pediatric Subjects With Type 1 Diabetes (TID)
Brief Title: Evaluation of Pharmacokinetics and Pharmacodynamic Properties of Rapid-Acting Insulin Analogs
Acronym: PK/PD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 403026582; JDRF Hypoglycemia Grant
Record Dates: First submitted 2008-03-27; First posted 2008-04-03 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus, Type I
Keywords: Type I Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro; Insulin Aspart; Insulin Detemir; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Catheter day 4 (Active Comparator): Adolescents with type 1 diabetes with catheters day #4
  Interventions: Drug: Insulin analogs (Lispro and Aspart)
- Catheter day 1 (Active Comparator): Adolescents with type 1 diabetes with catheter day #1
  Interventions: Drug: Insulin analogs (Lispro and Aspart)
- Aspart and Detemir (Active Comparator): Adolescents with type 1 diabetes
  Interventions: Drug: Insulin analogs (Aspart and Detemir)
- Lispro and Glargine (Active Comparator): Adolescents with type 1 diabetes
  Interventions: Drug: Insulin analogs (Lispro and Glargine)

INTERVENTIONS:
Drug: Insulin analogs (Lispro and Aspart) — Insulin bolus given through insulin pump
  Other Names: Humalog, Novolog
  Arms: Catheter day 1; Catheter day 4
Drug: Insulin analogs (Aspart and Detemir) — Drugs given separately
  Arms: Aspart and Detemir
Drug: Insulin analogs (Aspart and Detemir) — Drugs given in the same injection
  Arms: Aspart and Detemir
Drug: Insulin analogs (Lispro and Glargine) — Drugs given separately
  Arms: Lispro and Glargine
Drug: Insulin analogs (Lispro and Glargine) — Drugs given in single injection
  Arms: Lispro and Glargine

SUMMARY:
The aim of this study is to evaluate the variations in pharmacokinetic and pharmacodynamic properties of rapid-acting insulin analogs when given as a bolus by subcutaneous insulin infusion pump as typically encountered in the care of children with type 1 diabetes.

The specific factors under investigation are:

* the effects of puberty
* type of insulin analog
* site of catheter insertion
* and age of catheter

DETAILED DESCRIPTION:
The aim of this study is to evaluate the variations in pharmacokinetic (as determined by serum free insulin concentrations) and pharmacodynamic (as determined by the glucose infusion rate required to maintain euglycemia during a euglycemic clamp) properties of the rapid acting insulin analogs when given as a bolus by subcutaneous insulin infusion pump as typically encountered in the care of children with type 1 diabetes. The specific factors we will investigate are the effects of puberty (pre- vs. pubertal), type of insulin analog (lispro or aspart insulin), site of catheter insertion (gluteal vs. abdominal), and age of catheter (fresh insertion vs. three-day duration) Our hypotheses are that the peak (Imax) and area under the curve (IAUC) serum free insulin concentration, and the peak glucose infusion rate required to maintain euglycemia (GIRmax) and area under the curve (GIRAUC) will vary based on these conditions, in children given the same weight-based dose.

We will also evaluate the pharmacokinetic and pharmacodynamic properties of Aspart and Lispro insulin when used in a basal-bolus regimen with insulin Detemir or Glargine, new basal insulin analogs, given as separate injections and when combined in a single injection in adolescent patients with Type 1 DM. We hypothesize that the peak (IMAX) and area under the curve (IAUC) serum insulin concentrations, and the peak glucose infusion rate required to maintain euglycemia (GIRMAX) and area under the curve (GIRAUC) of the Aspart/Lispro bolus, will be similar when the Aspart/Lispro is combined in the same syringe with the insulin Detemir/Glargine, compared to when the Aspart/Lispro and Detemir/Glargine are given as two separate injections.

ELIGIBILITY:
Inclusion Criteria:

1. Age 8-17 (inclusive), of whom 15 will be prepubertal and 60 pubertal;
2. Clinical diagnosis of T1D (based on clinical presentation, insulin dependence,and/or history of ketosis;
3. Diagnosis of T1D for at least one year's duration;
4. On CSII therapy for at least three months;
5. HbA1c 6.5-8.0%, inclusive;
6. Body mass index < 95% for age and gender;
7. Meeting minimum weight requirement of at least 17.6 kg (for pre-pubertal subjects) or 34.6 kg (for pubertal subjects)
8. Ability to comprehend written and spoken English

Exclusion Criteria:

1. Any other medical disease aside from T1D or treated hypothyroidism
2. Receiving any other medication besides insulin or levothyroxine
3. Female subjects of reproductive potential who may be pregnant, breast feeding, or not consistently utilizing barrier methods or abstinence as contraception
4. Inability to comprehend written and spoken English
5. Any other condition, which in the judgement of the investigators, would interfere with the subject's or parents' ability to provide informed consent or the investigator's ability to perform the study

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2007-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Maximum Glucose Infusion Rate (GIR) to maintain euglycemia | Six hour observation period

SECONDARY OUTCOMES:
Time to Maximum Glucose Infusion Rate | Six Hour Observation period

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A Weinzimer, MD, Principal Investigator — Yale University; Eda Cengiz, MD, Principal Investigator — Yale University

REFERENCES:
- [Result] Cengiz E, Swan KL, Tamborlane WV, Sherr JL, Martin M, Weinzimer SA. The alteration of aspart insulin pharmacodynamics when mixed with detemir insulin. Diabetes Care. 2012 Apr;35(4):690-2. doi: 10.2337/dc11-0732. Epub 2012 Feb 28. PMID 22374642
- [Result] Cengiz E, Tamborlane WV, Martin-Fredericksen M, Dziura J, Weinzimer SA. Early pharmacokinetic and pharmacodynamic effects of mixing lispro with glargine insulin: results of glucose clamp studies in youth with type 1 diabetes. Diabetes Care. 2010 May;33(5):1009-12. doi: 10.2337/dc09-2118. Epub 2010 Feb 11. PMID 20150302
- [Result] Swan KL, Dziura JD, Steil GM, Voskanyan GR, Sikes KA, Steffen AT, Martin ML, Tamborlane WV, Weinzimer SA. Effect of age of infusion site and type of rapid-acting analog on pharmacodynamic parameters of insulin boluses in youth with type 1 diabetes receiving insulin pump therapy. Diabetes Care. 2009 Feb;32(2):240-4. doi: 10.2337/dc08-0595. Epub 2008 Nov 18. PMID 19017777
- [Result] Swan KL, Weinzimer SA, Dziura JD, Steil GM, Voskanyan GR, Steffen AT, Martin ML, Tamborlane WV. Effect of puberty on the pharmacodynamic and pharmacokinetic properties of insulin pump therapy in youth with type 1 diabetes. Diabetes Care. 2008 Jan;31(1):44-6. doi: 10.2337/dc07-0737. Epub 2007 Oct 1. No abstract available. PMID 17909083